CLINICAL TRIAL: NCT06630351
Title: Group Meaning-Centered Psychotherapy for Caregivers of Patients With Advanced Cancer
Brief Title: Group Meaning-Centered Psychotherapy for the Improvement of Wellbeing in Caregivers of Patients With Advanced Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deirdre R. Pachman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-004250; NCI-2024-07626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-004250 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-09-16; First posted 2024-10-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — Behavior Therapy; Health Promotion; Educational Status; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (MCP-C) (Experimental): Caregivers participate in MCP-C virtual group discussion sessions over 90 minutes each and complete reading exercises and workbook assignments once weekly for 8 weeks throughout the study.
  Interventions: Behavioral: Behavioral Counseling; Other: Discussion; Other: Health Promotion and Education; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Counseling — Participate in MCP-C
  Other Names: Behavior Counseling; Behavioral Psychotherapy
Other: Discussion — Participate in virtual group discussions
  Other Names: Discuss
Other: Health Promotion and Education — Receive reading exercises and workbook materials
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial assesses the acceptability and feasibility of a virtual group Meaning-Centered Psychotherapy for Cancer Caregivers (MCP-C) and its effect in improving the wellbeing of caregivers of patients with advanced cancer. Caregivers often suffer from significant existential distress, which includes feelings of hopelessness, demoralization, burden, loss of meaning and dignity, and a decreased will to live. MCP-C seeks to help caregivers connect to meaning and purpose despite the challenges of caregiving and helps caregivers understand how sources of meaning may help with symptoms of burden and reduce despair. Participating in MCP-C may help improve sense of personal meaning, spiritual well-being, and mood in caregivers of patients with advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine feasibility as measured by total number of caregivers enrolled in 1 year, adherence.

II. Determine acceptability as measured by satisfaction with the research process, as measured by the Was It Worth It (WiWi 2.0) questionnaire.

III. To evaluate preliminary efficacy of group MCP-C for personal meaning as measured by Life Attitude Profile-Revised (LAP-R), spiritual wellbeing as measured by Functional Assessment of Chronic Illness Therapy (FACIT) Spiritual Well-Being Scale (SWBS), depression and anxiety symptoms as measured by Hospital Anxiety and Depression Scale (HADS), meaning in caregiving as measured by Attitudes Towards Caregiving Scale (ATCS), social support as measured by Duke-University of North Carolina (UNC) Functional Social Support Questionnaire (FSSQ), benefit finding as measured by Benefit Finding Scale (BFS).

IV. Determine participants' perceptions of their experience with the intervention, including potential benefits they experienced, which components had the greatest impact, and whether they would suggest any changes to the intervention.

OUTLINE:

Caregivers participate in MCP-C virtual group discussion sessions over 90 minutes each and complete reading exercises and workbook assignments once weekly for 8 weeks throughout the study.

After completion of study intervention, caregivers are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* English fluency
* No diagnosed severe cognitive impairment
* Caregiver of a patient with diagnosis of advanced, solid tumor cancer (stage III/stage IV)
* Provide written (paper or electronic) informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Patient baseline distress score >= 4/10
* Have ability to utilize the technology to participate in virtual groups

Exclusion Criteria:

* As determined through self-report, those diagnosed with a history of a psychotic episode will be excluded
* Other psychological co-morbidities such as untreated schizophrenia, bipolar disease
* Cognitive impairment likely to interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Meaning-Centered Psychotherapy for Caregivers (MCP-C) intervention | Up to 1 year
  Feasibility will be measured by numbers and percentages of participant recruitment, enrollment, accrual, and retention of participants in the MCP-C intervention. Findings will be summarized using estimates and corresponding 95% confidence intervals.
Acceptability of MCP-C intervention | 4 months (2 months post intervention)
  Acceptability will be measured by the Was It Worth It (WIWI) Questionnaire. The WIWI consists of 7 questions, 3 answered with yes/no/uncertain, two answered on a 3-point scale (i.e., improved, stayed the same, or got worse), one open-ended/fill-in-the-blank question, and one yes/no question.

SECONDARY OUTCOMES:
Change in personal meaning - LAP-R | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  The Life Attitude Profile-Revised (LAP-R) is a 48-item scale that measures a person's life attitude and meaning in life. The LAP-R is scored on a 7-point Likert scale, with a minimum score of 30 and a maximum score of 210. A higher score indicates a greater sense of meaning in life and a more positive attitude towards life.
Change in spiritual well-being - FACIT-Sp-12 | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  Spiritual well-being will be assessed using the Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale (FACIT-Sp-12), a 12-item self-report measure with a total score range of 0-48, with higher scores indicating a greater level of spiritual well-being. items are answered on a scale of 0-4 where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, and 4=Very much.
Changes in anxiety and depression - HADS | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  Change in anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item self-rated questionnaire with depression and anxiety subscales both ranging from 0 to 21, categorized as: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Items are answered on a scale of 0-3 with varying responses for each question (e.g., very much/quite a lot/not very much/not at all or often/sometimes/not often/very seldom).
Change in attitude toward caregiving - ATCS | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  Change in attitude toward caregiving will be assessed using the Attitudes Towards Caregiving Scale ( ATCS), a 43-item 5-point Likert-type measure of ways caregivers find meaning through caregiving. The ATCS yields an overall (range 43-215) and three subscale [loss/powerlessness (range 19-96), provisional meaning (range 19-96), and ultimate meaning (range 5-25)] scores, with higher scores indicating higher overall meaning. Items are answered with one of 5 responses: strongly agree, agree, undecided, disagree, or strongly disagree.
Change in perception of social support - Duke-UNC FSSQ | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  Change in perception of social support will be assessed using the Duke/University of North Caroling (UNC) Functional Social Support Questionnaire (FSSQ), an 8-item measure of social support that generates a total score (range 0-44). Higher scores generally indicate a higher degree of satisfaction related to social support. Items are answered on a scale of 5-1 where 5=as much as I would like; 4=almost as much as I would like; 3=some, but would like more; 2=less than i would like, and 1=much less than I would like.
Change in benefit-finding - BFS | Baseline, 8 weeks (post intervention), 4 months (2 months post intervention)
  Change in perception of benefit will be assessed using the Benefit Finding Scale (BFS), a 17-item measure of perceived benefits adapted from Behr's Positive Contributions Scale for breast cancer, modified for caregiving. It yields a total score (range 17-85) with higher scores indicating greater benefit finding. Items are answered with one of 5 responses: not at all, a little bit, somewhat, quite a bit, or very much.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre R. Pachman, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials